CLINICAL TRIAL: NCT00074737
Title: Open Label, Phase II Dosing Study of Ara-C Chemotherapy in Combination With EL625 and Idarubicin in Refractory and Relapsed Acute Myelogenous Leukemia (AML)
Brief Title: Dosing Study of Ara-C/EL625/Idarubicin in Refractory and Relapsed AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eleos, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELP1001; 2003-0475 (MD Anderson)
Record Dates: First submitted 2003-12-19; First posted 2003-12-23 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Refractory or Relapsed Acute Myelogenous Leukemia (AML); Antisense
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — cenersen; OL(1)p53; Idarubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- cenersen, idarubicin (Active Comparator): cenersen, idarubicin, no cytarabine
  Interventions: Drug: cenersen; Drug: Idarubicin
- cenersen, idarubicin, cytarabine (Active Comparator): cenersen, idarubicin, standard dose cytarabine
  Interventions: Drug: cenersen; Drug: Idarubicin; Drug: Cytarabine
- cenersen, idarubicin, HDAC (Active Comparator): cenersen, idarubicin, HDAC (high dose cytarabine)
  Interventions: Drug: cenersen; Drug: Idarubicin; Drug: Cytarabine

INTERVENTIONS:
Drug: cenersen — cenersen with standard of care
  Other Names: cenersen sodium; Ol(1)p53; EL625; Aezea
Drug: Idarubicin — standard of care for AML
  Other Names: idamycin
Drug: Cytarabine — standard of care Ara-C and High dose Ara-C
  Other Names: Ara-C; HDAC
  Arms: cenersen, idarubicin, HDAC; cenersen, idarubicin, cytarabine

SUMMARY:
The principal goal of this clinical trial is to assess the ability of cenersen sodium (EL625) to improve cancer responsiveness to the established AML therapeutic agent Idarubicin used alone or in combination with Cytarabine (Ara-C).

Cenersen sodium is a drug that is designed to block the effects of a protein called p53. Laboratory evidence shows that blocking p53 will make many types of cancer, including acute myelogenous leukemia (AML), more sensitive to a variety of established cancer therapeutics while making normal tissues more resistant to the toxic effects of these agents.

DETAILED DESCRIPTION:
This clinical trial is designed to assess the ability of cenersen sodium (EL625) in combination with Idarubicin alone or with Cytarabine to either: (1) induce remissions in patients who have previously failed to go into remission in response to chemotherapy; or (2) provide patents who have relapsed after going into a chemotherapy-induced remission with a longer remission.

Cenersen sodium is one of a new class of drugs called antisense oligonucleotides (oligos). Oligos are designed to block the production of specific proteins and thereby inhibit their function. Cenersen sodium targets p53, a widely studied protein.

In cancer, p53 occurs either in the un-mutated ("normal") or mutated forms. The majority of participants in this trial are expected to have un-mutated p53. Cenersen sodium is anticipated to sensitize cancers with un-mutated p53 to most established cancer therapeutics.

p53 has a pivotal role in protecting the body from cells that have suffered genetic damage and, as a result, do not function properly. The protein first senses the level of the damage and then forces the damaged cell to respond to the damage either by repairing itself or committing suicide. In general, the greater the level of damage the more likely the cellular response will be suicide.

Many cancer therapeutics, including both chemotherapy and radiation, cause the types of genetic damage that activate p53 and, consequently, cause either damage repair or cellular suicide. Laboratory studies suggest that cancer cells have a host of defenses that reduce the chances that these cells will respond to genetic damage by committing suicide. So compared to normal cells, cancer cells are more likely to repair the damage caused by cancer therapeutics while normal cells are more likely to commit suicide. Thus, blocking un-mutated p53 is more likely to prevent repair in cancer cells while preventing suicide in normal cells. This provides the basis for a differential effect of cenersen sodium on cancer cells verses normal cells.

When p53-dependent repair is prevented in cancer cells they begin to copy their damaged genetic information in preparation for cell division. This copying of the genetic damage triggers a p53-independent backup suicide mechanism and, as a result, the cancer cells are eliminated. This is the presumed mechanism whereby cenersen sodium is able to sensitize cancer cells with normal p53 function to numerous cancer therapeutics.

At higher doses however, chemotherapy sometimes blocks cells from copying their genes in preparation for division. Thus, it is possible that a chemotherapeutic agent used at a high dose could block any sensitizing effect that cenersen sodium might otherwise have on the cancer.

The chemotherapeutic agent Idarubicin is known to produce the type of genetic damage that effects p53 expression, causes p53-dependent responses and has been shown to be made more effective at killing cancer cells by cenersen sodium. Cytarabine (Ara-C) is the most widely used chemotherapeutic agent for AML. Cenersen sodium does not appear to sensitize cancer cells to Cytarabine and at higher doses Cytarabine may reduce the capacity of cenersen sodium to sensitize cancer cells.

Hence, this AML study will examine the effects of Cenersen sodium used in combination with Idarubicin and one of three different doses of Cytarabine (i.e. 0, 0.1 and 1.0 gm/m2/day), on the responsiveness of participants to these chemotherapeutic agents.

ELIGIBILITY:
Inclusion Criteria

* Subjects with either refractory AML (not achieving a CR after a single course of induction), or relapsed AML that have a CR for less than one year.
* greater or equal to 18 years old.
* Life expectancy of more than 4 weeks following initiation of treatment.
* Performance status (Zubrod) less or equal to 3.
* Total Bilirubin less or equal to 1.5 x upper normal limit (UNL) unless attributable to organ infiltration by leukemia, and ALT(SGPT) less or equal to 2.5 x UNL.
* Creatinine less or equal to 1.5 x UNL unless attributable to organ infiltration by leukemia.
* If plasma creatinine value is borderline, creatinine clearance greater or equal to 60 ml/min (actual or calculated), serum magnesium should be within the normal value.
* Subjects with liver and/or renal dysfunction due to organ infiltration by leukemia are eligible.
* Left Ventricular Ejection Volume (LVEF) of >50% as determined by multi-gated acquisition scan (MUGA) or echocardiogram.
* Able to comply with scheduled follow-up and with management of toxicity.
* Sexually active patients must use an effective method of contraception during the study dosing period. The following are considered acceptable methods of contraception: (i) oral contraceptive pill, (ii) condom, (iii) diaphragm plus spermicide, (iv) patient or partner surgically sterile, (v) patient or partner more than 2 years post-menopausal or (vi) injectable or implantable agent/device.
* Informed consent form obtained, signed and dated prior to initiation of treatment

Exclusion Criteria:

* Subjects with M3 AML.
* Subjects receiving other anti-leukemia investigational agents (i.e., unapproved drugs). However, individual cases will be considered on a case-by-case basis for other investigational agents (e.g., antibiotics, antifungals).
* Pregnant or lactating subjects. Chemotherapy (including hydroxyurea) within three (3) weeks prior to initiation of therapy, unless there is evidence of rapidly progressive disease; then subjects may be enrolled with a minimum of two (2) weeks from previous treatments.

Prohibited Medications during the first week of each course:

* Acetaminophen
* Hi-Dose antioxidants (e.g., Vitamins C, E; Multivitamins)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2004-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Determine the effective dose of Cytarabine chemotherapy to be used in combination with EL625 and Idarubicin. | 6 months
  Cenersen plus standard of care

SECONDARY OUTCOMES:
Determine the safety profile for the combination of EL625 and Idarubicin +/- Cytarabine. | 6 months
  Standard of care plus cenersen
Determine the Complete Response Rate and Time to Progression. | 6 months
  Standard of care plus cenersen

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center; Edward D. Ball, MD, Principal Investigator — University of California, San Diego; John DiPersio, MD, Principal Investigator — Washington University Medical Center, Siteman Cancer Center; Maria Baer, Principal Investigator — Roswell Park Cancer Institute; Jonathan Kolitz, MD, FACP, Principal Investigator — North Shore University Hospital; Hugo Fernandez, MD, Principal Investigator — University of Miami
Locations (6):
- United States (6):
  - University of California, San Diego, La Jolla, California
  - University of Miami Health Center, Miami, Florida
  - Washington University Medical Center (Siteman Cancer Center), St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Lake Success, New York
  - M. D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: M.D. Anderson Cancer Center's website — http://www.mdanderson.org
- See also: University of Miami Medical Center — http://www.med.miami.edu/
- See also: Roswell Park Cancer Institute — http://www.roswellpark.org
- See also: Moores Cancer Center — http://cancer.ucsd.edu
- See also: Washington University Sch0ool of Medicine — http://medschool.wustl.edu